CLINICAL TRIAL: NCT00005360
Title: HIV Diversity and Pathogenesis in Donor-Recipient Clusters
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4247; R01HL048367 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2001-12

CONDITIONS: Acquired Immunodeficiency Syndrome; Blood Transfusion; Blood Donors; HIV Infections
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections

SUMMARY:
To assess, in donor-recipient clusters, current models of HIV-1 genetic evolution and pathogenesis, based on the sequence diversity displayed by this lentivirus.

DETAILED DESCRIPTION:
DESIGN NARRATIVE:

Based on anti-HIV-1 screening of a repository of 200,000 blood donor sera collected in late 1984, the Transfusion Safety Study identified and enrolled into ongoing followup 133 seropositive donors and 111 HIV-1-infected transfusion recipients. Included among these were 38 'transmission clusters' composed of a donor and from one to six linked, infected recipient(s), and, in four cases, infected recipients' sexual partners. Frozen cells and sera collected at six-month intervals over a six-year period from members of these clusters were available for study. Specimens were accessed such that sub-repositories of cellular DNA, PCR-amplified HIV-1 sequences, and viral isolates were generated for future investigations of these unique clusters. The studies included analysis of sequence diversity in envelope (env) V3, V4, and V5 hypervariable regions both within each infected individual over time, and between different members of each cluster and different clusters. Sequence diversity profiles from PBMC and serum were analyzed separately to discern differences in these different blood components at each sampling and over time. The pattern of turnover of specific sequence variants over time (evolution of viral genotypes) was correlated with clinical and immunological progression.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1992-08; Study Completion 1997-07 (Actual)

REFERENCES:
- [Background] Asher M. Plantar release in the correction of deformities of the foot in childhood. J Bone Joint Surg Am. 1982 Jun;64(5):790-1. No abstract available. PMID 7085708
- [Background] Diaz RS, Zhang L, Busch MP, Mosley JW, Mayer A. Divergence of HIV-1 quasispecies in an epidemiologic cluster. AIDS. 1997 Mar 15;11(4):415-22. doi: 10.1097/00002030-199704000-00003. PMID 9084787
- [Background] Sabino EC, Delwart E, Lee TH, Mayer A, Mullins JI, Busch MP. Identification of low-level contamination of blood as basis for detection of human immunodeficiency virus (HIV) DNA in anti-HIV-negative specimens. J Acquir Immune Defic Syndr (1988). 1994 Aug;7(8):853-9. PMID 8021818